CLINICAL TRIAL: NCT01044108
Title: A Randomized, Double-Blind, Placebo-Controlled, Two Part Trial (Sequential Single Subcutaneous Dose Rising Trial and Semi-Sequential Multiple Subcutaneous Dose Response Trial) to Investigate the Safety, Tolerability, Efficacy and Pharmacokinetics of NNC 0070-0002-0453 in Overweight/Obese Male and Female Subjects
Brief Title: A Two Part Trial Investigating an Anti-obesity Drug in Overweight/Obese Male and Female Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9161-3749; U1111-1112-7351 (Other: WHO)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial, part 1 (males only) (Experimental)
  Interventions: Drug: NNC 0070-0002-0453; Drug: placebo
- Trial, part 2 (males and females) (Experimental)
  Interventions: Drug: '2-0453; Drug: placebo

INTERVENTIONS:
Drug: NNC 0070-0002-0453 — Administration of a single subcutaneous (under the skin) dose. Up to 7 escalating dose levels will be investigated. Progression to next dose level will be based on a safety evaluation.
  Arms: Trial, part 1 (males only)
Drug: '2-0453 — Administration of multiple subcutaneous (under the skin) doses for 10 weeks. Up to 4 escalating dose levels will be investigated. Progression to next dose level will be based on a safety evaluation.
  Arms: Trial, part 2 (males and females)
Drug: placebo — Placebo will be administered as a comparator at each dose level.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate the safety, tolerability, efficacy and pharmacokinetics (the rate at which the trial drug is eliminated from the body) of NNC 0070-0002-0453 in overweight/obese, but otherwise healthy male and female volunteers. Selected subjects will continue in a follow-up period of up to 5 years.

DETAILED DESCRIPTION:
Due to an unfavourable benefit-risk profile observed during the phase 1 trial for the obesity project, NN9161, Novo Nordisk has decided to terminate further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* FOR TRIAL PART 1, THE FOLLOWING APPLIES:
* Informed consent must be obtained before any trial-related activities. Trial-related activities are any procedures that would not have been performed during the normal management of the subject
* Overweight/obese males: Body Mass Index (BMI) between 27.0 to 39.0 kg/m2
* Good general health
* FOR TRIAL PART 2, THE FOLLOWING APPLIES:
* Informed consent must be obtained before any trial-related activities. Trial-related activities are any procedures that would not have been performed during the normal management of the subject.
* Obese male and female subjects: Body Mass Index (BMI) between 30.0 to 39.0 kg/m2
* Good general health.

Exclusion Criteria:

* Aggressive diet attempts within the last 3 months
* Current or history of treatment with medications that may cause significant weight gain
* History of major depressive disorder or history of a suicide attempt or history of any suicidal behaviour
* History of eating disorders
* Any weight change of 5 kg (11 pounds) in the last 3 months
* Tobacco use
* History of alcoholism or drug/chemical abuse

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2011-09-20 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events | From the first trial related activity (Day 1) and until completion of the post treatment follow-up visit (Day 22 +/- 1)

SECONDARY OUTCOMES:
Terminal half-life (t½) | After administration of a single dose of trial drug
AUC 0-24h, area under the '2-453 concentration-time curve | From 0 to 24 hours after steady state

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Evansville, Indiana, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com